CLINICAL TRIAL: NCT06016829
Title: The Effect of Preoperative Nutritional Status, Dietary Inflammatory Index and Systemic Inflammatory Response on Postoperative Outcomes in Colorectal Cancer.
Brief Title: Preoperative Nutritional Status and Postoperative Outcomes in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Tuba Nur Yildiz Kopuz, Principal Investigator, Hacettepe University
Other Study IDs: GO 21/499
Record Dates: First submitted 2023-08-23; First posted 2023-08-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; nutritional status; body composition; quality of life; postoperative complication
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nutrition Risk Screening 2002 (NRS-2002) — Nutritional status assessment tool
Diagnostic Test: Global Leadership Initiative on Malnutrition (GLIM) — Nutritional status assessment tool
Other: Measurement of body composition with computed tomography (CT) — The cross section of the third lumbar vertebrae in the CT scan images of the patients will be analyzed for assessment of body composition parameters including skeletal muscle area (SMA), visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT)
Diagnostic Test: Dietary inflammatory index (DII) — The Dietary Inflammatory Index (DII) is a scoring algorithm that indicates the inflammatory potential of the diet.
Diagnostic Test: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) — Quality of life assessment tool
Diagnostic Test: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Colorectal Cancer 29 (EORTC-QLQ-CR29) — Quality of life assessment tool
Diagnostic Test: Prognostic Nutritional Index (PNI) — Prognostic Nutritional Index is diagnostic test based on serum albumin level and total lymphocyte count
Diagnostic Test: Neutrophil-Lymphocyte Ratio (NLR) — The neutrophil-to-lymphocyte ratio (NLR) is calculated as the simple ratio between neutrophil and lymphocyte counts.

SUMMARY:
The aim of this study was to evaluate the effect of preoperative nutritional status, dietary inflammatory index, and systemic inflammatory response on postoperative outcomes. The study will include 120 colorectal cancer patients who are scheduled for surgical treatment.

DETAILED DESCRIPTION:
A questionnaire form containing general information, dietary habits, and food consumption records will be applied by the researcher in the preoperative period to the patients who volunteered to participate in the study. Body composition will be taken by bioelectrical impedance analysis method. Hand grip strength will be taken with a digital hand dynamometer. The nutritional status of patients will be assessed using the criteria of the Nutritional Risk Screening 2002 (NRS-2002) and the Global Leadership Initiative on Malnutrition (GLIM). For body composition analysis, computed tomography images, known as the gold standard, will be used in cancer patients. Computed tomography images of the patients will be obtained from hospital records at L3 lumbar vertebra level. The software program ImageJ developed by the US National Institute of Health will be used to calculate the visceral fat area (cm2), subcutaneous fat area (cm2), and skeletal muscle area (cm2) from the recorded images.

Preoperative biochemical parameters will be obtained from hospital records. The systemic inflammatory response will be determined by the Prognostic Nutritional Index, Neutrophil Lymphocyte Ratio, and Delta Neutrophil Index. The inflammatory load of the diet will be calculated using the Dietary Inflammatory Index. The quality of life of patients will be assessed using cancer-specific scales developed by the European Organisation for Research and Treatment of Cancer (EORTC) during the preoperative and postoperative periods. These scales are EORTC-QLQ-C30 for general quality of life and EORTC-QLQ-CR29 for colorectal cancer-specific quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with colorectal cancer and having surgical treatment planned
* Being 18 years of age or older

Exclusion Criteria:

* Having received chemotherapy or radiotherapy
* Currently undergoing corticosteroid or hormone treatment.
* Presence of distant metastases.
* Presence of any malignancy other than colorectal cancer.
* Presence of autoimmune disease.
* Presence of ongoing infectious disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who have undergone surgical treatment for a diagnosis of colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | within 30 days after surgery
  Complications graded by Clavien-Dindo Complication Classification System
Postoperative quality of life | within 45 days after surgery
  Quality of life will be evaluated by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30).All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
EORTC-QLQ-CR29 | within 45 days after surgery
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Colorectal Cancer 29 (EORTC-QLQ-CR29) is a supplementary questionnaire module to be employed in conjunction with the Quality of Life Questionnaire Core 30 (QLQ-C30). All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scale and functional single-items represents a high level of functioning, whereas a high score for the symptom scales and symptom single-items represents a high level of symptomatology or problem.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba N Yildiz Kopuz, Principal Investigator — Hacettepe University; Mehmet Fisunoglu, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Ankara
  - Ankara City Hospital Bilkent, Ankara